CLINICAL TRIAL: NCT02942797
Title: Nutritional Risk Screening 2002 Should be Used to Predict Prognostic Outcomes in Chronic Obstructive Pulmonary Disease With Respiratory Failure
Brief Title: NRS 2002 as a Predictor of Prognosis in COPD With Respiratory Failure
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lu Xing, Principal Investigator, Master Degree, West China Hospital
Other Study IDs: COPD-002
Record Dates: First submitted 2016-10-11; First posted 2016-10-24 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NRS 2002 score ≥ 3
- NRS 2002 score < 3

SUMMARY:
This is a prospective study of patients diagnosed with chronic obstructive pulmonary disease (COPD) with respiratory failure and admitted in West China Hospital during April 2017 to March 2019. The following variables will be prospectively studied: age, sex, height, weight, respiratory function indicators, arterial blood gas analysis results, biochemical data, nutritional risk screening 2002 (NRS 2002) score, short-term and long-term prognostic outcomes. The purpose of this study is to assess whether NRS 2002 is a useful prognosis predictor in COPD patients with respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosis of COPD at West China Hospital during April 2017 to March 2019
* Partial pressure of O2 (PaO2) < 60 mmHg and/or partial pressure of CO2 (PaCO2) >50 mmHg
* Age ≥ 18 years
* Respiratory rates > 23 bpm

Exclusion Criteria:

* Pregnancy or during lactation
* Ventilatory dysfunction due to neuromuscular disorders, acute and chronic thromboembolic disease, severe illness in other systems
* Refused to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with chronic obstructive pulmonary disease with respiratory failure during April 2017 to March 2019 at West China Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Predictive value of NRS 2002 in identifying COPD patients with respiratory failure who will have poor prognostic outcomes, in terms of mortality | up to 2 years
Predictive value of NRS 2002 in identifying COPD patients with respiratory failure who will have poor prognostic outcomes, in terms of 30-day readmission after discharge | up to 2 years
Predictive value of NRS 2002 in identifying COPD patients with respiratory failure who will have poor prognostic outcomes, in terms of length of stay | up to 2 years
Predictive value of NRS 2002 in identifying COPD patients with respiratory failure who will have poor prognostic outcomes, in terms of complications | up to 2 years

SECONDARY OUTCOMES:
Collection of Demographics (age, sex) | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China